CLINICAL TRIAL: NCT04183114
Title: Immunogenicity & Safety of Bio Farma's Measles-Rubella (MR) Vaccine in Indonesian Infants (Bridging Study)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MR-BF 0319
Record Dates: First submitted 2019-08-28; First posted 2019-12-03 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Congenital Rubella Infection; Measles
Keywords: Vaccine; Measles; Rubella; Bio Farma
MeSH Terms: conditions — Measles; Rubella

STUDY DESIGN:
Intervention Model Description: healthy infants aged 9 - 12 months
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking uses observer blind with some unmasked staff to prepare the vaccine to be administered by masked investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IP batch MRUK-0317 (Experimental): 135 Subjects received Bio Farma's vaccine batch MRUK 0317
  Interventions: Biological: Measles-Rubella vaccine Bio Farma
- IP Batch MRUK-0417 (Experimental): 135 Subjects received Bio Farma's vaccine batch MRUK 0417
  Interventions: Biological: Measles-Rubella vaccine Bio Farma
- IP Batch 550118 (Experimental): 135 Subjects received Bio Farma's vaccine batch MRUK 0417
  Interventions: Biological: Measles-Rubella vaccine Bio Farma
- Control (Active Comparator): 135 Subjects received SII's MR vaccine batch 012W72230Z
  Interventions: Biological: MR Vaccine SII

INTERVENTIONS:
Biological: Measles-Rubella vaccine Bio Farma — MR vaccine produced by Bio Frama with 3 consecutive batches
  Other Names: Vaksin Campak Rubella Bio Farma
  Arms: IP Batch 550118; IP Batch MRUK-0417; IP batch MRUK-0317
Biological: MR Vaccine SII — MR Vaccine produced by SII (Already registered in Indonesia)
  Arms: Control

SUMMARY:
Thus study is a clinical trial for Measles and Rubella vaccine that will be used inIndonesian National Program of Immunization. The study design will be randomized, observer blind, prospective intervention study.

DETAILED DESCRIPTION:
The objectives of the study are:

* To assess the protectivity rate of Bio Farma's Measles/Rubella (MR) vaccine in infants
* To describe antibody response to Measles and Rubella after 1 dose of Bio Farma's MR vaccine as a primary dose in infants
* To assess the safety of Bio Farma's Measles/Rubella (MR) vaccine in infants
* To evaluate immunogenicity and safety one dose of Bio Farma's MR vaccine compare to registered MR vaccine.
* To evaluate immunogenicity and safety in three consecutive batches of Bio Farma's MR vaccine in infants .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Infants, 9-12 months
2. Parents have been informed properly regarding the study and signed the informed consent form
3. Parents will commit themselves to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial.
2. Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature > 37.5 Centigrade).
3. Known history of allergy to neomycin, kanamycin or erythromycin or any component of the vaccines.
4. History of immunodeficiency disorder or disorders like HIV infection, leukemia, lymphoma, or generalized malignancy that can alter immune response.
5. Subjects who have previously received any measles and/or rubella containing vaccines.
6. Subjects who had a clinical history of measles/rubella infection.
7. Subjects who has received in the previous 3 months a treatment likely to alter the immune response (intravenous immunoglobulin, blood-derived products or long term corticosteroidtherapy (> 2 weeks).
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
9. Subject already immunized with any vaccine within 4 weeks prior vaccination.

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Protectivity of Measles | 4 months
  Percentage of subjects with anti measles titer ≥ 8(1/dil), 28 days after one dose of Bio Farma's MR vaccine in Infants
Protectivity of Rubella | 4 months
  Percentage of subjects with anti rubella titer ≥11 IU/ml, 28 days after one dose of Bio Farma's MR vaccine in Infants

SECONDARY OUTCOMES:
Immunogenicity of MR Vaccine in infants GMT | up to 4 months
  • Serological response to MR vaccine in infants: GMT
Immunogenicity of MR Vaccine (4 Folds increase of antibody titer) | up to 4 months
  • Serological response to MR vaccine in infants: percentage of infants with increasing antibody titer > 4 times.
Immunogenicity of MR Vaccine (seroconversion) | up to 4 months
  • Serological response to MR vaccine in infants: percentage of infants with transition of seronegative to seropositive.
Comparison Between MR (Bio Farma) Vaccine and Registered MR Vaccine | up to 4 months
  • Comparability of serological response to Measles and Rubella component, pre and post vaccination with Bio Farma's MR vaccine compared to registered MR vaccine in infants.
Comparison between each batch number of Bio Farma's MR vaccine. | up to 4 months
  • Serological response between each batch number of Bio Farma's MR vaccine.
Safety (immediate reactions) | up to 30 minutes after vaccination
  • Immediate reactions within the first 30 minutes after vaccination
Safety (72 hours) | up to 72 hours after vaccination
  • Local reactions and systemic events occurring within 72 h after vaccination.
Safety (14 days) | up to 14 days after vaccination
  • Local reactions and systemic events occurring within 14 days after vaccination
Safety (15 days to 28 days) | up to 14 days
  • Local reactions and systemic events occurring between 15 days to 28 days following injection.
Safety (Serious adverse event) | up to 1 months/28 days
  • Any serious adverse event occurring from inclusion until 28 days after immunization
Safety comparison between MR vaccine and control | up to 1 months/28 days
  • Description of adverse events between MR vaccine and control.
Safety comparison between each batch of MR vaccine | up to 1 months/28 days
  • Description of adverse events between each batch number of MR vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Child Health Dept. Dr. Soetomo Hospital, School of Medicine Airlangga Univ., Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
no plan for IPD. Data are restricted to be used by investigators and sponsor only.